CLINICAL TRIAL: NCT07405827
Title: Prospective Follow-up Study of Patients Undergoing Shoulder Instability Surgery
Brief Title: French Shoulder Instability Surgery Cohort Study
Acronym: ShoulderCDS
Status: Recruiting | Type: Observational
Sponsor: Chirurgie Du Sport (Other)
Responsible Party: Principal Investigator, HARDY Alexandre, Surgeon, Chirurgie Du Sport
Other Study IDs: ShoulderCDS
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Shoulder Instability Subluxation Bilateral; Shoulder Instability
Keywords: shoulder; instability; bankart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Shoulder instability surgery — Shoulder instability surgery encompasses procedures aimed at restoring stability to the glenohumeral joint following recurrent dislocations or subluxations.
  Bankart repair (anterior or posterior) involves reattaching the detached labrum to the glenoid rim and tightening the associated capsulolabral structures to restore joint stability.
  Latarjet (Butée) procedure consists of transferring the coracoid process with its attached muscles to the anterior glenoid, providing a bony and dynamic restraint to prevent recurrent dislocations.
  These procedures aim to restore joint stability, improve functional outcomes, and enable safe return to sport. They are selected based on the type, direction, and severity of instability, as well as patient-specific factors.
  Other Names: Bankart repair (anterior/posterior); Latarjet (Butée)

SUMMARY:
This 20-year cohort study follows patients after shoulder instability surgery to evaluate recurrence rates, long-term functional outcomes, return-to-sport rates, and complications.

The goal is to provide insights into the durability and effectiveness of surgical treatment in order to improve patient care.

DETAILED DESCRIPTION:
This study is a long-term cohort analysis involving patients who have undergone shoulder instability surgery. The goal is to follow these patients over a 20-year period to assess several important outcomes. Specifically, the study aims to evaluate the rate of recurrence, the rates and quality of return to sport, long-term functional outcomes using validated scoring systems, and the incidence of complications related to the procedure.

By collecting detailed and consistent data over two decades, the research seeks to provide valuable insights into the durability and effectiveness of surgical treatment for shoulder instability, contributing to a better understanding and improved care for patients.

ELIGIBILITY:
Inclusion Criteria

Patients undergoing surgical treatment for shoulder instability, including:

Bankart repair (anterior or posterior) Latarjet (Butée) procedure

Exclusion Criteria Patient refusal

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients enrolled in the ShoulderCDS cohort by one of the surgeons of the Chirurgie du Sport and meeting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2042-04-30 (Estimated); Study Completion 2062-04-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of dislocation or subluxation of the operated shoulder | From the surgery to the end of the study (20years of follow-up for each patient)

SECONDARY OUTCOMES:
Return to sport | From the surgey to the end of follow up (20 years)
  Return to sport after surgery with the level of return, the type of sport and the delay. Questions regarding the return to sport at 6 months, 1 year, 2 years and every 2 years
Shoulder Instability Surgery - Return to Sport Injury score | From the surgery to the end of follow-up (20 years for each patient).
  The SIRSI (Shoulder Instability - Return to Sport Injury) score is used to assess the patient's psychological readiness and apprehension regarding their return to sport following surgical stabilization of the shoulder. The score ranges from 0% (lowest level of psychological readiness) to 100% (highest level of psychological readiness). Questionnaires are administered at 6 months, 1 year, 2 years, and every 2 years thereafter.
Western Ontario Shoulder Instability Index (WOSI) | From the surgery to the end of follow-up (20 years per patient).
  The WOSI (Western Ontario Shoulder Instability Index) is a validated patient-reported outcome measure used to assess shoulder function, pain, and quality of life in patients with shoulder instability. It consists of multiple domains, including physical symptoms, sports/recreation, lifestyle, and emotions. Scores range from 0 to 2100, with higher scores indicating worse shoulder-related quality of life. Questionnaires are administered at 6 months, 1 year, 2 years, and every 2 years thereafter to monitor long-term functional outcomes.
Walch-Duplay Score | From the surgery to the end of follow-up (20 years per patient).
  The Walch-Duplay score is a clinician-administered assessment used to evaluate functional outcomes and stability of the shoulder after surgical stabilization. It includes domains for pain, stability, range of motion, and ability to perform sports or daily activities. Scores range from 0 to 100, with higher scores indicating better shoulder function and stability. Assessments are performed at 6 months, 1 year, 2 years, and every 2 years thereafter to monitor long-term recovery and functional outcomes.
ROWE score | From the surgery to the end of follow-up (20 years per patient).
  The Rowe score is a clinician-administered assessment used to evaluate shoulder stability, function, and pain following surgical treatment for shoulder instability. It includes components for stability, motion, and functional ability, with a total score ranging from 0 to 100, where higher scores indicate better shoulder function and stability. Assessments are performed at 6 months, 1 year, 2 years, and every 2 years thereafter to monitor long-term outcomes.
Visual Analogue Scale | From the surgery to the three day after surgery
  The VAS score (Visual Analogue Scale) is a simple and widely used method for assessing subjective experiences, such as pain intensity, fatigue, or discomfort. It typically consists of a horizontal or vertical line, usually 10 cm in length, with endpoints representing the extremes of the experience being measured: 0: "No pain" (or "no discomfort"). 10: "Worst pain imaginable" (or "maximum discomfort") Evaluated during the 3 first days after surgery
Complications | From the surgery to the end of follow-up (20 years per patient).
  Complications of the surgery and any re-operations will be recorded, including:
  Removal of hardware Infection Hematoma Revision shoulder stabilization Cartilage surgery Arthrodesis Shoulder prosthesis

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Hardy, MD, Principal Investigator — Chirurgie Du Sport
Locations (1):
- Chirurgie du Sport, Paris, Île-de-France Region, France